CLINICAL TRIAL: NCT06452316
Title: An Open-Label Study Evaluating the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Subjects With Limbal Stem Cell Deficiency
Brief Title: Study to Evaluate the Safety and Efficacy of CSB-001 Ophthalmic Solution 0.1% in Subjects With Limbal Stem Cell Deficiency
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Claris Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSB-C23-001
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Observation (non-interventional) for 20 weeks followed by one drop CSB-001 four times daily for two 8-week dosing periods in the study eye(s) separated by >30 days and <40 days followed by observation (non-interventional) for 52 weeks (total participation of 96 weeks)
  Interventions: Biological: CSB-001 Ophthalmic Solution 0.1%
- CSB-001 QID (Experimental): One drop CSB-001 four times daily for two 8-week dosing periods in the study eye(s) separated by >30 days and <40 days followed by observation (non-interventional) for 72 weeks (total participation of 96 weeks)
  Interventions: Biological: CSB-001 Ophthalmic Solution 0.1%

INTERVENTIONS:
Biological: CSB-001 Ophthalmic Solution 0.1% — CSB-001: human recombinant dHGF (5-amino acid deleted hepatocyte growth factor)

SUMMARY:
This study will enroll subjects with qualifying limbal stem cell deficiency (LSCD). All subjects will receive CSB-001 investigational drug in either one or both study eyes. The study is comprised of two identical phases (Dosing Phase I and II) of test article dosing separated by a 31- to 40-day period, the Dosing Holiday, where no test article is administered. Dosing Phase II is followed by an observational, noninterventional phase (Observation Phase).

ELIGIBILITY:
Inclusion Criteria:

* Have an area of the central 5 mm zone of cornea affected, presence of at least one clinical sign observed by slit-lamp examination with white light and/or cobalt blue light, fluorescein, and a Wratten filter, and at least one clinical sign observed with AS-OCT.
* If dosing with Acthar at time of Screening Visit, must have a history of stable dosing for approximately 8 weeks, plan to maintain the same Acthar treatment dose and regimen, and have demonstrated little to no improvement in severity of LSCD.
* Sponsor written confirmation of qualifying LSCD diagnosis.
* Inflammation associated with LSCD or other non-infectious inflammation that will not interfere with subject's participation.

Exclusion Criteria:

* Any active ocular infection (bacterial, viral, fungal, or protozoan) in either eye.
* Ocular surgery within 30 days of Day 0 where investigator assesses that healing is not considered complete/stable.
* Planned ocular surgery on or before Week 20 visit.
* Presence or history of any ocular or systemic disorder, condition, or procedure that might hinder the efficacy of the study treatment or its evaluation, or could interfere with the interpretation of study results, in the opinion of the investigator.

Note: Other inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety as Assessed by Adverse Event Reporting | Day 0 through Week 96
  Incidence of ocular and systemic adverse events
Safety as Assessed by Slit-lamp Biomicroscopy | Day 0 through Week 96
  Change from baseline in slit-lamp parameters
Safety as Assessed by Best-corrected Distance LogMAR Visual Acuity | Day 0 through Week 96
  Change from baseline using the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart

SECONDARY OUTCOMES:
Efficacy as Assessed by Change in Stage of LSCD | Day 0 through Week 96
  Change from baseline in LSCD signs based on imaging (white light, blue light with fluorescein and Wratten filter, and AS-OCT)
Efficacy as Assessed by Change in Best-corrected Distance LogMAR Visual Acuity | Day 0 through Week 96
  Visual acuity measured using the EDTRS visual acuity chart

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Loma Linda University Eye Institute, Loma Linda, California
  - Midwest Cornea Associates, LLC, Carmel, Indiana
  - Francis Price Jr, MD, Indianapolis, Indiana
  - Minnesota Eye Consultants, Minnetonka, Minnesota
  - Legacy Devers Eye Institute, Portland, Oregon
  - Stuart A. Terry, MD PA, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No